CLINICAL TRIAL: NCT06755463
Title: The Effect of Acupressure on Beta-Endorphin, Hypocretin, Cognition, and Patient-Reported Outcome Measures in Multiple Sclerosis Patients (APEX-MS Trial): a Single-Blind, Randomized Controlled Trial
Brief Title: Acupressure in MS Patients
Acronym: APEX-MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-HSF-SDEMIR-05
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; pain; fatigue; cognition; quality of life; depression
MeSH Terms: conditions — Multiple Sclerosis; Pain; Fatigue; Depression

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-blind, randomized, controlled, and experimental trial. It involves two parallel groups: an intervention group and a control group.
  Participants in the intervention group will receive acupressure therapy for 8 weeks, applied twice per week, following structured training provided by a certified practitioner. The therapy targets specific acupressure points associated with pain relief, fatigue reduction, cognitive improvement, and emotional regulation.
  Participants in the control group will receive routine clinical care without any acupressure intervention during the study period. However, they will be trained in acupressure techniques and provided educational materials at the end of the study.
Who Masked: Outcomes Assessor
Masking Description: In this clinical trial, the outcome assessors are masked to the group assignments to minimize evaluation bias. Participants are not masked, as those in the intervention group will receive acupressure therapy, while the control group will receive routine care without acupressure. Data analysts will receive de-identified data for analysis to further reduce bias during statistical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will receive acupressure therapy for 8 weeks, with twice-weekly sessions between 8:00 AM and 10:00 AM. A certified practitioner will train them on acupressure principles, including target points, pressure techniques, frequency, and duration. Practical demonstrations will ensure correct technique application. Training groups of up to 10 participants will learn the method in a comfortable setting. The protocol targets beta-endorphin and hypocretin levels, cognition, and patient-reported outcomes (pain, fatigue, depression, and quality of life). 6 acupressure points (LI4, SP6, GV20, HT7, EX-HN3, and LV3) will be used, totaling 12 symmetrical points. Pressure will be applied for 2 minutes per point using 3-5 kg force in rhythmic movements, totaling 24 minutes. Participants will practice under supervision, receive a diary to track home practice, and be given a visual guide for proper technique.
  Interventions: Other: Self-acupressure education
- Control group (No Intervention): Participants in the control group will not receive any acupressure therapy during the study period. They will continue to receive routine clinical care as recommended by their physicians. After the study concludes, acupressure points and techniques will be demonstrated and taught to participants in this group. They will also receive the same visual guide/brochure provided to the intervention group, explaining each acupressure point and application method in detail.

INTERVENTIONS:
Other: Self-acupressure education — Participants will undergo acupressure therapy for 8 weeks, with twice-weekly sessions between 8:00 AM and 10:00 AM. A certified practitioner will train participants on target points, pressure techniques, frequency, and duration. Practical demonstrations will ensure correct application. Groups of up to 10 participants will be trained in a comfortable setting and practice techniques under supervision until proficient. The treatment protocol, based on literature, focuses on beta-endorphin and hypocretin levels, cognition, and patient-reported outcomes (pain, fatigue, depression, and quality of life). Participants will apply 3-5 kg pressure for 2 minutes per point at 12 symmetrical points (LI4, SP6, GV20, HT7, EX-HN3, LV3) using rhythmic movements, totaling 24 minutes. They will receive a diary to track home practices and a visual guide explaining each point's location and steps for application.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effects of acupressure therapy on patients with Multiple Sclerosis (MS). MS is a chronic autoimmune disease affecting the central nervous system, characterized by inflammation, demyelination, and nerve damage. Patients often experience symptoms such as fatigue, muscle weakness, pain, depression, anxiety, and cognitive impairment, which lower their quality of life and make daily activities challenging. In addition to conventional treatments, complementary therapies can help alleviate these symptoms. Acupressure is a non-invasive technique that involves applying pressure to specific points on the body to regulate energy flow, without using needles.

This research investigates the effects of acupressure on beta-endorphin and hypocretin levels, cognitive functions, and patient-reported symptoms in MS patients. Beta-endorphin is known as a natural pain reliever, while hypocretin plays a role in regulating sleep-wake cycles and energy levels. The study hypothesizes that acupressure can increase the levels of these biochemical substances, improving pain, fatigue, and cognitive functions.

This single-blind, randomized controlled trial will include 82 MS patients. Participants will be divided into two groups: the intervention group (receiving acupressure therapy) and the control group (receiving routine care). The acupressure intervention will be performed twice a week for eight weeks. Participants in the intervention group will learn acupressure techniques and apply them as part of the treatment, while those in the control group will receive acupressure training after the study ends.

Throughout the study, beta-endorphin and hypocretin levels will be measured via blood tests, and cognition, pain, fatigue, depression, and quality of life will be assessed using validated scales. Participants will also report their experiences during the treatment, and the data collected will be analyzed through comparative evaluations.

This research aims to comprehensively analyze the effects of acupressure on MS patients and provide scientific evidence regarding the effectiveness of complementary therapies. The findings may offer an alternative method to improve quality of life and alleviate symptoms for MS patients. Acupressure's simplicity, affordability, and ease of application make it a more accessible and sustainable option. The study will be conducted in compliance with ethical standards, prioritizing participant safety.

DETAILED DESCRIPTION:
Background Multiple Sclerosis (MS) is a chronic autoimmune and neurodegenerative disease affecting the central nervous system (CNS). It is characterized by inflammation, demyelination, gliosis (scar formation), and axonal damage. These pathological changes lead to impairments in motor and cognitive functions, sensory perception, vision, and balance. The unpredictable progression of MS contributes to physical disability and psychological distress, significantly reducing patients' quality of life.

Current treatments primarily focus on disease-modifying therapies (DMTs) to slow disease progression and symptomatic management strategies to address pain, fatigue, depression, and cognitive impairments. However, conventional approaches often fail to fully alleviate symptoms, leading patients to seek complementary and alternative therapies. Acupressure has emerged as a promising complementary method due to its non-invasive, low-cost, and easy-to-apply nature.

Acupressure is based on Traditional Chinese Medicine principles and involves applying pressure to specific points on the body. It aims to balance energy flow and promote physiological and psychological well-being. Studies have demonstrated its effectiveness in reducing pain, fatigue, and stress and improving sleep quality and cognitive function. However, evidence on its impact on neuropeptides such as beta-endorphin and hypocretin in MS patients remains limited.

Beta-endorphin is an endogenous opioid peptide known for its analgesic properties, stress modulation, and role in emotional regulation. Hypocretin (also called orexin) regulates arousal, wakefulness, and energy balance. Dysregulation of these neuropeptides has been implicated in MS-related symptoms, including fatigue, pain, and cognitive decline. This study aims to explore whether acupressure can modulate these biomarkers and improve clinical outcomes in MS patients.

The APEX-MS study (Trial of Acupressure and Patient Experience in Multiple Sclerosis) aims to investigate the effects of acupressure on beta-endorphin levels, hypocretin levels, cognition, and patient-reported outcome measures (PROMs) in individuals with MS.

Methods This study will be conducted using a single-blind, randomized, controlled, and experimental design. The research will take place at the Neurology Clinic of Bolu Abant İzzet Baysal University İzzet Baysal Training and Research Hospital. The study population will consist of individuals who have been diagnosed with MS and followed up for at least six months. The sample size was determined using the GPower 3.1.9.7 software, and a total of 82 participants (41 in each group) were calculated to be sufficient for the study.

Participants will be randomly assigned to either the intervention group (receiving acupressure therapy) or the control group (receiving placebo intervention) using stratified randomization. Stratified randomization will ensure balanced distribution of key variables such as age, gender, disease severity, and disease duration. The randomization sequence will be generated by an independent researcher who is not involved in data collection or analysis.

As required by the single-blind design, researchers assessing outcomes, including beta-endorphin and hypocretin levels, cognitive functions, and PROMs, will remain unaware of group assignments. This approach will minimize evaluation bias and ensure reliable results.

Inclusion Criteria:

* Diagnosis of MS confirmed by a neurologist based on the McDonald criteria.
* Having the Relapsing-Remitting MS (RRMS) subtype.
* Diagnosed with MS for at least one year.
* Individuals aged between 18 and 65 years.
* Expanded Disability Status Scale (EDSS) score between 0 and 5 (indicating mild to moderate disability).
* No use of steroid treatment or discontinuation of steroid therapy at least 3 months prior to study participation.
* No MS relapse in the past 3 months.
* No prior use of acupressure or similar complementary therapies.
* Sufficient language proficiency to understand and complete study assessments and questionnaires.

Exclusion Criteria:

* Presence of any open wounds or deformities at the acupressure application site.
* Diagnosis of neurodegenerative or neuropsychiatric diseases such as - -
* Parkinson's or Alzheimer's, which may potentially confound study results.
* Pregnant or breastfeeding women, due to potential hormonal changes that may affect results.
* Presence of severe cardiovascular, pulmonary, hepatic, renal, or psychiatric conditions.

Hypotheses of the study:

H1-1: Acupressure increases beta-endorphin levels in MS patients, contributing to the alleviation of symptoms such as pain, fatigue, and stress.

H1-2: Acupressure regulates hypocretin levels in MS patients, leading to improvements in fatigue and cognitive functions.

H1-3: Acupressure enhances cognitive functions in MS patients, and this improvement is associated with changes in beta-endorphin and hypocretin levels.

H1-4: Acupressure improves PROMs, resulting in reduced pain and fatigue, decreased depression scores, and enhanced overall quality of life.

Data collect and measures As part of the study, individuals registered at the neurology outpatient clinic will first be screened using the hospital's database. During this screening process, eligibility will be assessed based on inclusion and exclusion criteria, including age (18-65 years), duration of diagnosis (at least one year), and the presence of additional diagnosed and monitored conditions (e.g., neurodegenerative and neuropsychiatric diseases). Information on eligible patients will be recorded in a list. Patients included in the list will be contacted by phone, and further assessments will be conducted based on the inclusion and exclusion criteria. The Expanded Disability Status Scale (EDSS) score (0-5 points) will be evaluated, along with the presence of steroid therapy, the time since the last MS relapse, pregnancy or breastfeeding status, and prior use of acupressure or similar complementary therapies. Patients will receive preliminary information about the study's purpose, goals, expected outcomes, and duration, and their willingness to participate voluntarily will be assessed. Patients who do not meet the criteria will be excluded from the list, while eligible patients will be invited to the hospital's outpatient clinic for the study initiation. Prior to the clinic visit, a randomization sequence will be generated, and participants will be assigned to either the intervention or control group. The study flow diagram is provided in Figure 1 for detailed reference. Upon arrival at the clinic, participants will be thoroughly informed about the study (its purpose, goals, responsibilities, and duration), and written informed consent will be obtained.

All participants in this study, regardless of group assignment, will first undergo data collection procedures to obtain baseline (Time-0/T0) measurements. A "Demographic and Clinical Information Form" will be administered at the start of the study to gather data on participants' age, gender, education level, employment status, disease duration, EDSS score, and the number of MS relapses experienced in the past year. The study will examine the measurement variables detailed below, and the corresponding data collection tools will be applied at the specified time points listed. All data will be collected through face-to-face interviews with participants. However, data on pain and fatigue measured at the T1 time point will be collected via telephone interviews.

Measurement variable-1: Laboratory Data (Beta-Endorphin and Hypocretin Levels) Data collection form: Laboratory Data Monitoring Form Description: Measurement of beta-endorphin and hypocretin levels will not require any additional blood sampling from participants as part of the study. The levels of these biomarkers will be obtained from blood samples collected during routine clinical follow-ups requested by the neurologist. Blood samples will be drawn via venous access into 2 ml biochemistry tubes as part of standard clinical procedures in the neurology department. No additional invasive procedures will be performed for this study. Beta-endorphin and hypocretin levels will be analyzed using specialized ELISA kits. Samples will be sent to an external laboratory following routine blood collection in the outpatient clinic. Reported results will be recorded in the monitoring form and used for the study's statistical analyses.

Measurement time points: T0 and T2.

Measurement Variable-2: Cognition Data Collection Tool: Brief International Cognitive Assessment for MS (BICAMS)

Description:

BICAMS is a test battery with strong psychometric properties, developed in 2012 to rapidly and effectively assess cognitive dysfunction in patients with MS. The Turkish version of this form was validated in 2017. BICAMS consists of three short tests that evaluate three key cognitive domains:

Symbol Digit Modalities Test (SDMT): This test includes a key table with symbols and corresponding numbers, along with a sequence of symbols. The key table shows which number corresponds to each symbol (e.g., a triangle corresponds to the number "3"). The participant is presented with the key table and a series of symbols underneath it. The participant is asked to write the correct number below each symbol by referring to the key table. Two methods are available for administration: written (pen-and-paper) and oral (verbal response). In this study, the oral method will be individually administered. The participant's score is based on the number of correct matches completed within 90 seconds. The SDMT measures information processing speed and attention, and the highest possible score is 110. The test takes approximately 5 minutes to complete.

California Verbal Learning Test, Second Edition (CVLT-II): CVLT-II is a standard measure of auditory/verbal learning and memory widely used in clinical neuropsychology. In this study, the first five trials assessing verbal memory will be used. The test consists of 16 words grouped into 4 categories (4 vehicles, 4 vegetables, 4 animals, and 4 pieces of furniture). CVLT-II evaluates not only the number of words recalled but also learning and recall strategies, including errors, repetitions (perseverations), and intrusions. The total correct recall across the five trials represents the learning score. The maximum possible score is 80.

Brief Visuospatial Memory Test Revised (BVMT-R): BVMT-R assesses visuospatial memory through three recall trials. The test consists of a stimulus card displaying six geometric figures arranged in a 2x3 grid. In each trial, participants are shown the card for 10 seconds and then asked to draw as many figures as possible in their correct positions on a blank sheet of paper. Each correctly drawn figure earns a maximum of two points, and the total score for all six figures across three trials is 36 points. The difference between the first and third trials is used to assess learning progress.

Measurement Time Points: T0 (Baseline) and T2 (Post-intervention).

Measurement variable-3: PROMs (pain, fatigue, depression, quality of life) Pain Severity Assessment: Pain severity will be evaluated using the Visual Analog Scale (VAS). The VAS consists of a 10 cm scale (0 = no pain, 10 = worst possible pain), where participants will mark the point that best represents their pain intensity (measured at time points: T0, T1, and T2).

Fatigue Assessment: Fatigue will be assessed using the Fatigue Severity Scale (FSS). This is a 9-item test that evaluates how fatigued participants have felt during the past week, including the day of assessment. Participants rate each item on a scale from 1 (strongly disagree) to 7 (strongly agree) based on their experience. The total score is divided by the number of items to calculate the average score. A score of 4 or higher typically indicates pathological fatigue. The Turkish validity and reliability study conducted by Armutlu et al. (2007) reported a Cronbach's alpha coefficient of 0.89 (measured at time points: T0, T1, and T2).

Depression Assessment: Depression levels will be evaluated using the Beck Depression Inventory (BDI). The BDI is a 21-item self-assessment scale designed to measure symptoms in vegetative, emotional, cognitive, and motivational domains. Participants will evaluate how they have felt over the past week, including the assessment day, by selecting the most suitable response for each item. Scores range from 0 to 3 for each item, with a total score range of 0-63. A total score of 17 or above is considered indicative of depression. The Turkish validity and reliability study reported a Cronbach's alpha coefficient of 0.80. This assessment will be conducted at time points: T0 and T2.

Quality of Life Assessment: Quality of life will be measured using the Multiple Sclerosis Impact Scale-29 (MSIS-29), developed by Hobart et al. in 2001. This tool includes 20 items related to physical parameters and 9 items covering psychological issues. Items 1-20 measure physical impact, while items 21-29 assess psychological impact. Participants are asked to rate how MS has affected their daily lives over the past two weeks using a 5-point Likert scale. Scores from the two subscales can be combined and converted to a scale of 0-100, with higher scores indicating greater disease impact. The Turkish validity and reliability study conducted by Özden et al. (2022) reported Cronbach's alpha coefficients of 0.968 for the physical domain and 0.914 for the psychological domain. This assessment will be conducted at time points: T0 and T2.

The study will consist of two groups: the intervention group and the control group. While the intervention group will receive acupressure therapy, the control group will receive no intervention and will continue with routine care. The specific interventions for each group are detailed below:

Intervention Group:

Participants in this group will undergo acupressure therapy for 8 weeks, receiving sessions twice a week between 8:00 AM and 10:00 AM. They will be trained by a certified acupressure practitioner on the fundamental principles of acupressure, including the target points, pressure techniques, frequency, and duration of application. Practical demonstrations will be provided to ensure participants understand the techniques.

On the day of their clinic visit, participants will be divided into groups of up to 10 people for training. The researcher will first ensure participants are in a comfortable position, then demonstrate the location and application methods for each acupressure point.

The treatment protocol, designed based on existing literature, focuses on evaluating the effects of acupressure on beta-endorphin and hypocretin levels, cognition, and patient-reported outcomes (pain, fatigue, depression, and quality of life).

Each acupressure point will be stimulated for 2 minutes using an average pressure of 3-5 kg, applied with the thumb, index finger, and/or middle finger in rhythmic movements synchronized with breathing. A total of 6 acupressure points have been identified for self-application: LI4 (Hegu), SP6 (Sanyinjiao), GV20 (Baihui), HT7 (Shenmen), EX-HN3 (Yin Tang), and LV3 (Tai Chong). With symmetrical points included, the total number of points will be 12.

LI4 (Hegu): Known for its analgesic effects and its ability to increase endorphin levels.

SP6 (Sanyinjiao): Promotes hormonal balance and general relaxation. GV20 (Baihui): Supports cognitive functions and brain performance. HT7 (Shenmen) and EX-HN3 (Yin Tang): Help alleviate depression symptoms, boost energy, and reduce fatigue.

LV3 (Tai Chong): Regulates energy flow, promotes balance, and enhances overall health.

The acupressure trainer will first apply pressure to each point for 2 minutes, totaling 24 minutes (120 seconds × 12 points = 1620 seconds = 24 minutes). Participants will then practice self-application under supervision until they are able to perform the technique correctly.

Participants will also be given an acupressure diary to track their home practice sessions and ensure compliance. Additionally, they will receive a visual guide/brochure explaining each acupressure point's location and step-by-step application instructions.

Control Group:

Participants in the control group will not receive any acupressure therapy during the study period. They will continue to receive routine clinical care as recommended by their physicians. After the study concludes, acupressure points and techniques will be demonstrated and taught to participants in this group. They will also receive the same visual guide/brochure provided to the intervention group, explaining each acupressure point and application method in detail.

Data Analysis and Reporting At the end of the 8-week study, all participants, regardless of group assignment, will be invited to the neurology outpatient clinic for a face-to-face evaluation. Blood samples collected during routine monitoring by a specialist neurologist to assess beta-endorphin and hypocretin levels will be sent to an external laboratory for analysis. At the T2 time point, participants will complete data collection tools through individual face-to-face interviews. Additionally, participants in the control group will receive training on acupressure techniques in groups of up to 10 people and will be provided with a brochure explaining acupressure methods. The collected data will be entered into a statistical analysis program and securely stored on the principal investigator's computer. The data analysis process will be conducted as follows: The Shapiro-Wilk test will be used to assess whether the data follows a normal distribution. Non-parametric tests will be employed for data that do not meet normality assumptions. Descriptive statistics, including mean, standard deviation, median, and range, will be calculated for participants' demographic characteristics (age, gender, MS type, etc.) and outcome measures. Pre-test and post-test comparisons between groups will be conducted using independent samples t-tests or Mann-Whitney U tests. Within-group comparisons will be analyzed using paired samples t-tests or the Wilcoxon Signed-Rank Test. If normality and assumptions are met, Analysis of Covariance (ANCOVA) will be applied to determine differences between the acupressure and control groups. ANCOVA will control for baseline values (covariates) to assess post-test differences between groups. For measurements taken at three time points, Repeated Measures ANOVA will be performed to evaluate time-dependent changes. Effect sizes, such as eta squared, will be calculated to determine the clinical relevance of observed changes over time. A p-value < 0.05 will be considered statistically significant. This approach ensures a comprehensive analysis of data to determine the effectiveness of acupressure on biochemical markers, cognition, and patient-reported outcomes in MS patients.

During the implementation of the study, all ethical principles will be strictly adhered to. Participants' personal information and health data will be protected in accordance with confidentiality principles and will only be accessible to authorized researchers. Approval for conducting the study was obtained from the administration of Bolu Abant İzzet Baysal University İzzet Baysal Training and Research Hospital, and ethical approval was granted by the Non-Interventional Clinical Research Ethics Committee.

Before the study begins, all participants will receive detailed information about the acupressure applications, potential risks, benefits, and the implementation process. Written informed consent will be obtained from each participant. Participants will be trained on identifying the correct acupressure points, applying appropriate pressure, and recognizing possible side effects. This training will be provided through face-to-face sessions by a certified acupressure practitioner who is an experienced nurse with theoretical and practical expertise.

Previous studies have demonstrated that acupressure is a safe method, with no adverse events reported to date. However, participants will be asked to report any side effects (e.g., pain, dizziness, nausea) experienced after each session in the Acupressure Diary specified in Appendix 6. These reports will be regularly reviewed, and participants will be able to contact researchers by phone if they experience any discomfort.

Participants will be clearly informed about conditions that may pose risks during acupressure application, such as pregnancy, severe skin diseases, bleeding disorders, or certain chronic illnesses, as well as contraindications like infected areas or open wounds. Individuals with such conditions will undergo necessary screenings and will not be included in the study.

Other safety measures will be ensured by clearly defining the inclusion and exclusion criteria of the study. No invasive procedures will be applied to participants, and there will be no risk of physical harm during the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an MS diagnosis confirmed by a neurologist based on the McDonald criteria.
* Having the RRMS subtype.
* Diagnosed with MS for at least one year.
* Individuals aged 18-65 years.
* An EDSS score between 0 and 5, indicating mild to moderate disability.
* No use of steroid therapy or discontinuation of steroid therapy at least 3 months prior to participation.
* No MS relapse within the last 3 months.
* No prior use of acupressure or other complementary therapies.
* Sufficient language proficiency to understand the study and complete assessments.

Exclusion Criteria:

* Presence of any open wounds or deformities at the application site.
* Presence of neurodegenerative or neuropsychiatric disorders such as - Parkinson's or Alzheimer's, which may potentially confound the study results.
* Pregnant or breastfeeding women, due to hormonal changes that may affect outcomes.
* Presence of severe cardiovascular, pulmonary, hepatic, renal, or psychiatric diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Beta-Endorphin levels | from baseline to two months
  Beta-endorphin levels will be measured using blood samples collected during routine clinical follow-ups, eliminating the need for additional invasive procedures. These biomarkers will be analyzed in an external laboratory using ELISA kits, and the results will be recorded and used for statistical analysis.
Hypocretin levels | from baseline to two months
  Hypocretin levels will be measured using blood samples collected during routine clinical follow-ups, eliminating the need for additional invasive procedures. These biomarkers will be analyzed in an external laboratory using ELISA kits, and the results will be recorded and used for statistical analysis.
Cognition | from baseline to two months
  Cognition in this study will be assessed using BICAMS, which includes SDMT for processing speed, CVLT-II for verbal memory, and BVMT-R for visual memory. These tests are validated tools for evaluating cognitive impairment in MS patients. Higher scores indicate better cognitive performance, and results will be analyzed to determine the impact of the intervention.

SECONDARY OUTCOMES:
Pain measurement | from baseline to two months
  Pain will be assessed using the VAS, a validated tool for measuring pain intensity. The scale ranges from 0 (no pain) to 10 (worst possible pain), with participants marking a point that best represents their pain level. Higher scores indicate greater pain severity. Results will be analyzed to evaluate changes in pain perception.
Fatigue | from baseline to two months
  Fatigue will be assessed using the FSS, a validated 9-item tool that evaluates the impact of fatigue on daily activities. Each item is scored from 1 (strongly disagree) to 7 (strongly agree). The total score is averaged, with higher scores indicating more severe fatigue. A score of 4 or above suggests clinically significant fatigue. Results will be analyzed to assess changes in fatigue levels.
Depression | from baseline to two months
  Depression will be assessed using the BDI, a validated 21-item self-report questionnaire measuring symptoms of depression. Each item is scored from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms. A score of 17 or above suggests clinically significant depression. Results will be analyzed to evaluate changes in depression levels.
Quality of life measurement | from baseline to two months
  Quality of Life will be assessed using the MSIS-29, a validated tool designed to measure the physical and psychological impact of MS. It consists of 20 items assessing physical health and 9 items evaluating psychological well-being. Each item is rated on a 5-point Likert scale, and total scores range from 0 to 100, with higher scores indicating a greater impact of the disease. Results will be analyzed to assess changes in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Seyma Demir Erbas, PhD, Principal Investigator — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: No
Participant confidentiality is ensured.